CLINICAL TRIAL: NCT00225914
Title: Paroxetine Controlled Release in the Treatment of Symptomatic Menopausal Women Following Discontinuation of Hormone Therapy
Brief Title: Study of Paxil Use in Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Lee S. Cohen, MD, Perinatal and Reproductive Psychiatry Program
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-P-000115
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Menopause
Keywords: Menopause; Hormone Therapy; Paxil; Hot Flash; Sleep Disturbance; Night Sweats; Antidepressants
MeSH Terms: conditions — Hot Flashes; Parasomnias | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects enter into a six-week, double blind phase, randomized in a 1:1 ratio to paroxetine CR 12.5 mg/day; dosing may be adjusted up to 25 mg/day after two weeks, based on treatment response and tolerability.
  Interventions: Drug: Paroxetine
- 2 (Placebo Comparator): Subjects then enter into a six-week, double blind phase, randomized in a 1:1 ratio to paroxetine CR 12.5 mg/day or matching placebo pill
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Paroxetine — Paroxetine CR 12.5 mg/day; dosing may be adjusted up to 25 mg/day after two weeks, based on treatment response and tolerability
  Other Names: Paxil
  Arms: 1
Drug: placebo — Subjects enter into a six-week, double blind phase, randomized in a 1:1 ratio to paroxetine CR 12.5 mg/day or matching placebo pill; dosing may be adjusted up to 25 mg/day after two weeks, based on treatment response and tolerability.
  Arms: 2

SUMMARY:
To evaluate the efficacy, safety, and tolerability of Paroxetine treatment in perimenopausal and postmenopausal women who present with menopause-related symptoms after discontinuing hormone therapy (HT), in the presence or absence of concomitant symptoms of depression or anxiety.

DETAILED DESCRIPTION:
This study is a 10-week double-blinded treatment study of perimenopausal and postmenopausal women who present with menopause-related symptoms after discontinuing Hormone Therapy(HT), with or without concomitant symptoms of depression and anxiety.

The menopausal transition is a period of heightened vulnerability to mood and anxiety disturbances. It is also a period when women may experience significant vasomotor symptoms (i.e. hot flushes and night sweats). More recently, the occurrence of vasomotor symptoms has been associated with increased risk for depression in menopausal women.

The efficacy of estrogens for the treatment of vasomotor symptoms is well established. In addition, the literature support a modulatory effect exerted by estrogen on various neurotransmitter systems that regulate mood and anxiety.

Despite the efficacy of hormone therapy (HT) for the treatment of menopause-related symptoms, a significant number of women discontinue its use during the first year of treatment. Moreover, recent findings from the Women's Health Initiative Study (WHI) have challenged the safety and the benefits that were initially thought to be associated with long-term use of HT. As a result, many women who have been taking HT decided to discontinue the use of HT, which may result in significant changes in their physical well being, quality of life and, possibly, their mental health status. Therefore, the efficacy and tolerability of other interventions such as antidepressants for these sub-populations warrant further investigation.

Treatment with Paroxetine has shown to be efficacious for menopause-related vasomotor symptoms. To date, no studies have examined the extent to which SSRIs may improve physical and psychological symptoms in women who discontinued HT.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 40 and above.
2. Perimenopausal status (defined as having cycles which vary by more than 7 days from normal, or 2 or more skipped cycles and an amenorrheic interval of at least 60 days but no more than 12 consecutive months) or postmenopausal status (defined as amenorrheic for 12 or more consecutive months).
3. Women with prior use of HT for at least two months.
4. Women who discontinued HT use 1 to 12 months prior to study entry (screening visit).
5. Women who present with significant menopause-related symptoms (defined as GCS total score >20; vasomotor sub-scores >3 and/or ³14 moderate to severe hot flashes per week), with or without concomitant psychological complaints (symptoms of depression and/or anxiety).
6. Women who report physical/emotional symptoms developing or worsening within 3 months of HT discontinuation.
7. General good health.

Exclusion Criteria:

1. Women who present with moderate-to-severe symptoms of depression (MADRS scores > 19) or anxiety (BAI scores > 19) at baseline.
2. Women who meet diagnostic criteria at screening visit for a current major Axis I psychiatric disorder other than specific phobias (assessed through M.I.N.I. interview). Subjects presenting with symptoms of anxiety or depression, but not meeting criteria for Depressive Disorders, Bipolar Disorder, Panic Disorder, GAD, OCD or SAD, will be allowed in the study.
3. Regular treatment with hormonal medications, SSRIs, tricyclic antidepressant, mood stabilizer, oral neuroleptics, sedatives or hypnotics, over-the-counter agents known to influence hot flushes or mood within 4 weeks prior to screening visit; used of depot neuroleptics within 12 weeks prior to screening visit.
4. Suicidal ideation, homicidal ideation, or psychotic symptoms.
5. Menstrual dysfunction and amenorrhea of other etiologies.
6. History of seizure disorder
7. Pregnancy or breastfeeding.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Mean change from Visit 2 to Visit 4 in the daily hot flash frequency and severity. Response will be considered if ³50% reduction in the hot flash composite score-frequency X severity) | 6 weeks

SECONDARY OUTCOMES:
Proportion of subjects with remission of menopause-related symptoms from Visit 2 to Visit 4 measured by a >50% decrease in Greene Climacteric Scale total and sub-scores and Hot Flush Related Daily Interference Scale (HFRDIS). | 6 weeks
Occurrence of discontinuation symptoms (DESS- Discontinuation Emergent Signs Symptoms, self-report) at Visit 4. | 6 weeks
Proportion of CGI responders (clinician-rated CGI- Improvement 2; Occurrence of adverse events (PRISE-Adverse Event Visit Checklist) throughout the study | 8 weeks
Proportion of subjects with remission of psychological symptoms (MADRS <10; BAI < 11 at Visit 4). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee S. Cohen, M.D., Principal Investigator — MGH Center for Perinatal and Women's Mental Health
Locations (1):
- MGH Center for Perinatal and Women's Mental Health, Boston, Massachusetts, United States

REFERENCES:
- See also: MGH Center for Perinatal and Women's Mental Health — http://www.womensmentalhealth.org